CLINICAL TRIAL: NCT02552472
Title: Haphazard and Careless Use of Inhalers, an Observational Study
Brief Title: A Study of Inhaler Use in the Community
Status: Completed | Type: Observational
Sponsor: Beaumont Hospital (Other)
Collaborators: Asthma Society Ireland (Unknown); Irish Thoracic Society (Other); GlaxoSmithKline (Industry); Vitalograph Ireland (Unknown); Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor Richard W Costello, Beaumont Hospital
Other Study IDs: INCA-CC
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Airways Disease
Keywords: Asthma; Inhaler Use; Adherence; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective cohort observational study of inhaler adherence in a community care setting (ie. general practice clinics and pharmacies in the community).

DETAILED DESCRIPTION:
Over a 2-4 week period, consecutive patients with a history of respiratory illness already prescribed a salmeterol/fluticasone Diskus inhaler will be asked to participate in this study. Patients will give informed consent to participate in this study of adherence, which will be assessed with the INCA device. Both clinicians and patients will be fully aware that the device is an acoustic recording device and that both time and technique of inhaler use will be assessed. Once consented, patients will be given an INCA enabled inhaler for 1 month and asked to use it as they normally would and then to return it at the end of one month. The days used and the number of doses used in the study period, as per the dose counter, will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Known history of Respiratory Illness
* Prescribed salmeterol/fluticasone Diskus Inhaler

Exclusion Criteria:

* Unable to understand study protocol
* Refusal to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a random sample of patients with a known history of respiratory illness and already prescribed a salmeterol/fluticosone Diskus inhaler. Patients will be identified in both community pharmacy centres and general practice clinics within Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Inhaler Adherence in Time | One month
  This is adherence as measured by the INCA device in regards to time of use. This is measured as a rate of use.
Inhaler Technique Adherence | One Month
  This is adherence measured by the INCA device in regards to technique of use. This is measured as a rate.

SECONDARY OUTCOMES:
Age Measured in Years at time of recruitment | one month
  Relationship of Age to Adherence
Gender Measured as Male or Female | One Month
  Relationship of Gender to Adherence
Education Level Measured as either primary, secondary or tertiary school at recruitment. | One Month
  Relationship of Education Level (Primary/Secondary/Tertiary) to Adherence
Socio-economic Class Measured as the patient having either Private or Public Health Insurance | One Month
  Relationship of Socio-economic class (Private or Public Health Insurance) to Adherence
Health Care Use Measured as the number of visits to a General Practitioner in the previous Year | Previous Year
  Relationship of Health Care Use (Frequency of visit to General Practitioner) to Adherence
Hospitalisation Measured as the number of hospital admissions in the previous year | Previous Year
  Relationship of Hospitalisation in the prevoius year to Adherence
Exacerbation Measured as the number of Respiratory Related Exacerbations in the previous year | Previous Year
  Relationship of Exacerbation (Respiratory related in the prevoius year) to Adherence
Background Respiratory Diagnosis, divided into Asthma, COPD and other. | Previous History
  Relationship of Respiratory Diagnosis (Asthma, COPD, other) to Adherence
Smoking History measured by three categories: 1. Current Smoker, 2. Ex-Smoker and 3. Never Smoker | Previous History
  Relationship of Smoking History (Current, Ex-smoker, never smoker) to Adherence

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, MD, Principal Investigator — RCSI, Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Dublin, Ireland